CLINICAL TRIAL: NCT02347813
Title: Chemoprevention of Squamous Cell Cancer of the Skin in High Risk Patients
Brief Title: Preventing Squamous Cell Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Alice Pentland, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: URochester RSRB 00052209
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-02

CONDITIONS: Squamous Cell Carcinoma of the Skin
Keywords: squamous cell carcinoma; pioglitazone; PPARgamma; skin cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carotid Intimal Medial Thickness 1; Skin Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delayed Intervention (Other): After enrollment, subjects will be observed for 24 weeks for skin cancer tumors. Tumors will be appropriately treated as per standard of care. Then they will begin the pioglitazone regimen for 24 more weeks, during which time skin cancer tumors will be observed and appropriately treated as per standard of care.
  Interventions: Drug: Pioglitazone
- Immediate Intervention (Other): Subjects will begin the 24 week pioglitazone regimen immediately after enrollment, during which time skin cancer tumors will be observed and appropriately treated as per standard of care. After 24 weeks of drug, subjects will be observed for 24 weeks for skin cancer tumors. Tumors will be appropriately treated as per standard of care.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 15 mg of pioglitazone orally for 2 weeks, and if well tolerated, 30 mg pioglitazone orally for 5 1/2 months.
  Other Names: Actos

SUMMARY:
This study is proposed based on our work showing that the diabetes drug Pioglitazone strongly inhibits growth of tissue cultured squamous cell carcinoma (SCC) of the skin. This occurs at concentrations readily achievable by oral administration of this drug using doses currently approved for the treatment of diabetes. In our study, we propose to enroll 40 non-diabetic adult subjects (18-80 yrs of age inclusive) with a documented clinical history of frequent occurrence of skin squamous cell cancer to receive Pioglitazone (Actos®,Takeda Pharmaceuticals). Each subject will receive usual care for all new tumors they develop while on study (i.e, excision and plastic repair). The study protocol will randomize (1:1) patients for 6 months of observation followed by 6 months of treatment (group 1) or 6 months of treatment with drug followed by observation for 6 months (to examine washout effects). The biopsy specimens collected on and off therapy will be examined to determine if they express AKR1C3, an enzyme we believe increases resistance of SCC to prostaglandin inflammatory mediators. We will also examine the histologic grade of the removed tumors and study whether Pioglitazone treatment can decrease the number of aggressive versus well differentiated tumors in study patients. This pilot study is designed to detect a statistically significant change in SCC tumor numbers but is not sponsored by the drug manufacturer. The data obtained will not be used to effect a change in the product label.

DETAILED DESCRIPTION:
This is a single center open label feasibility pilot project based at the University of Rochester. This study is proposed based on our work showing that the diabetes drug Pioglitazone strongly inhibits growth of tissue cultured squamous cell carcinoma (SCC) of the skin. This occurs at concentrations readily achievable by oral administration of this drug using doses currently approved for the treatment of diabetes. In our study, we propose to enroll 40 non-diabetic adult subjects (18-80 yrs of age inclusive) with a documented clinical history of frequent occurrence of skin squamous cell cancer to receive Pioglitazone (Actos®,Takeda Pharmaceuticals). Patients followed in the University of Rochester Dermatology Clinic who have had greater than 3 or more SCCs treated in the past year, without contraindication for the use of pioglitazone, and are on a stable drug treatment regimen will be offered participation .The study has a cross-over design, so patients will be enrolled and randomized to one arm of two treatment protocols: 1) six months of usual care while documenting and characterizing any new tumors that occur followed by 6 months of pioglitazone treatment plus usual care for the next 6 months or 2) six months of pioglitazone treatment followed by 6 months off treatment receiving usual care. The second group will offer the opportunity to assess whether there is any persistent beneficial effect after pioglitazone treatment ends, while tumors from the first group that occur during the initial 6 months of usual care will be characterized by study parameters for comparison to tumors arising while on treatment. At the end of the one year treatment period, the number of biopsy-proven new tumors that patients develop while taking pioglitazone will be counted and compared with the number that patients developed during the 6 month period they were not receiving treatment as well as the numbers that occurred during the 6 months after treatment (washout effect). This information will be used as the basis for a larger multicenter study. We will also examine the histologic grade of the removed tumors and study whether Pioglitazone treatment can decrease the number of aggressive versus well differentiated tumors in study patients. This pilot study is designed to detect a statistically significant change in SCC tumor numbers but is not sponsored by the drug manufacturer. The data obtained will not be used to effect a change in the product label.

This study will also assess secondary endpoints. First, we will examine whether the ratio of well-differentiated to poorly differentiated SCC is influenced while subjects are on treatment. This endpoint is included because it is unknown whether there may be more signaling mediated by PPARγ in one tumor morphology vs. another. Second, we will determine whether patients on treatment might have different numbers of "borderline" lesions biopsied; precancerous lesions are often suspicious enough to biopsy. It may be that there will be fewer lesions in this category, as well as fewer squamous cell cancers. Basal cell cancers and other forms of skin cancer will also be documented. Third, we will test tumors that are excised after they are processed for routine diagnostic pathology to see if markers of proliferation or apoptosis that are influenced by PPARγ activity or the presence of AKR1C3 are altered. These endpoints would support the idea that any changes produced in tumor incidence while patients are on study drug are related to the mechanistic effect on PPARγ that is proposed.

Subjects will be excluded from study if they have NYHA class I - IV cardiac status because of concerns that thiazolidinediones, such as Pioglitazone, may exacerbate congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age, male or female, state of health stable
* Able understand protocol and give consent
* Has had treatment of 2 - 6 squamous cell carcinomas of the skin during the year prior to enrollment, & pathology is available for verification
* Stable treatment regimen for their skin cancer problems in place for 1 year, with expectation to keep medications the same during study
* Able to keep study appointments & comply with protocol

Exclusion Criteria:

* Unwillingness or unable to complete informed consent process
* < 18 years of age
* Allergy to Pioglitazone
* Taking Rifampin, Trimethoprim, Celebrex or Gemfibrozil
* Pregnant or breastfeeding (Pregnancy Category C)
* History of heart failure NYHA Class III or Class IV
* Subjects with type 1 or type 2 diabetes
* Problems with pedal edema
* Liver disease (ETOH, viral hepatitis, drug-induced hepatitis) or elevated ALT, AST or total bilirubin
* Osteoporosis with high risk of fracture
* History of bladder cancer
* Recent change in chronic oral medications. Participants enrolled while on a systemic medication for their skin cancer must remain on treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P. Pentland, M.D., Principal Investigator — University of Rochester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mantel A, Carpenter-Mendini A, VanBuskirk J, Pentland AP. Aldo-keto reductase 1C3 is overexpressed in skin squamous cell carcinoma (SCC) and affects SCC growth via prostaglandin metabolism. Exp Dermatol. 2014 Aug;23(8):573-8. doi: 10.1111/exd.12468. Epub 2014 Jul 16. PMID 24917395

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirteen subjects consented, 1 subject screen failed, 2 subjects from the Delayed Intervention Arm were Early Terminations, 2 subjects from the Immediate Intervention Arm were Early Terminations, resulting in 4 subjects being randomized in to the Delayed Intervention Arm and 4 subjects being randomized in to the Immediate Intervention arm.
Groups:
- No Intervention, Then Pioglitazone: After enrollment, subjects will be observed for 24 weeks for skin cancer tumors. Tumors will be appropriately treated as per standard of care. Then they will begin the pioglitazone regimen for 24 more weeks, during which time skin cancer tumors will be observed and appropriately treated as per standard of care. There was no washout period.
  Pioglitazone: 15 mg of pioglitazone orally for 2 weeks, and if well tolerated, 30 mg pioglitazone orally for 5 1/2 months.
- Pioglitazone, Then no Intervention: Subjects will begin the 24 week pioglitazone regimen immediately after enrollment, during which time skin cancer tumors will be observed and appropriately treated as per standard of care. After 24 weeks of drug, subjects will be observed for 24 weeks for skin cancer tumors. Tumors will be appropriately treated as per standard of care. There was no washout period.
  Pioglitazone: 15 mg of pioglitazone orally for 2 weeks, and if well tolerated, 30 mg pioglitazone orally for 5 1/2 months.
Period: First Intervention, 24 Weeks
Arm/Group | No Intervention, Then Pioglitazone | Pioglitazone, Then no Intervention
Started | 6 | 6
Completed | 4 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Second Intervention, 24 Weeks
Arm/Group | No Intervention, Then Pioglitazone | Pioglitazone, Then no Intervention
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention, Then Pioglitazone | Pioglitazone, Then no Intervention | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Squamous Cell Carcinomas
Description: Squamous Cell Carcinomas were counted by visual inspection of the all skin on the body.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: # of squamous cell carcinomas
Groups:
- No Intervention: Standard of care
Arm/Group | No Intervention | Pioglitazone
Number analyzed (Participants) | 8 | 8
# of squamous cell carcinomas | 0.75 (0.71) | 1.00 (1.31)
Statistical Analysis 1: Comparison: No Intervention vs Pioglitazone; Test type: Other; p = 0.750, ANOVA; Mean Difference (Final Values) = 0.50

2. Secondary Outcome: Mean Number of Other Skin Cancers
Description: Cancers were counted by visual inspection of the all skin on the body. Patients were inspected for the following cancer types: squamous cell carcinoma, basal cell carcinoma and melanoma.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: # of other carcinomas
Arm/Group | No Intervention | Pioglitazone
Number analyzed (Participants) | 8 | 8
# of other carcinomas | 1 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | No Intervention | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=12) | Pioglitazone (N=12)
Metastatic squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=12) | Pioglitazone (N=12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was under enrolled and therefore was not powered to show a difference between the two arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02347813/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02347813/Prot_SAP_001.pdf